CLINICAL TRIAL: NCT02498431
Title: Serum Irisin Levels in Myocardial Infraction and Following Percutaneous Coronary Intevention
Brief Title: Serum Irisin in Myocardial Infraction and Following Percutaneous Coronary Intevention
Acronym: IRICARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 424 General Military Hospital (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Consultant of Endocrinology, 424 General Military Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRICARDIO
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: irisin; myocardial infarction; coronary
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Angioplasty, Balloon; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- myocardial infraction (Experimental): Patients with acute myocardial infraction who are admitted to the emergency department of 424 General Military Hospital before and after percutaneous coronary intervention and stent placement
  Interventions: Procedure: percutaneous coronary intervention; Procedure: coronary angiography; Device: Stent, Medronic Resolute Integrity
- coronary artery disease (Active Comparator): Patients with coronary artery disease but not myocardial infraction who are being subjected to coronary angiography and percutaneous coronary intervention and stent placement
  Interventions: Procedure: percutaneous coronary intervention; Procedure: coronary angiography; Device: Stent, Medronic Resolute Integrity
- Control (Active Comparator): Patients subjected to coronary angiography and found with no presence of coronary artery disease
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: percutaneous coronary intervention — a non-surgical procedure used to treat the stenotic (narrowed) coronary arteries of the heart found in coronary heart disease
  Other Names: coronary angioplasty
  Arms: coronary artery disease; myocardial infraction
Procedure: coronary angiography — is a procedure performed along with cardiac catheterization that uses X-ray imaging to see your heart's blood vessels
Device: Stent, Medronic Resolute Integrity — A stent is placed in an artery as part of a procedure called percutaneous coronary intervention (PCI) to restore blood flow through narrow or blocked arteries. A stent helps support the inner wall of the artery in the months or years after PCI.
  Arms: coronary artery disease; myocardial infraction

SUMMARY:
The investigators aim to evaluate circulating irisin levels alterations in patients with acute myocardial infraction and in patients with coronary artery disease subjected to percutaneous coronary intervention.

DETAILED DESCRIPTION:
Irisin is a newly discovered myokine induced in exercise. There is evidence that cardiac muscle produces more irisin than skeletal muscle in response to exercise. Furthermore, irisin has been associated with isoproterenol-induced myocardial infarction (MI) in rats while it has been reported to decrease after acute myocardial infarction in humans.

The investigators aim 1) to investigate circulating irisin levels in patients at the time of acute myocardial infarction and after reprefusion [primary percutaneous coronary intervention (PCI)] 2) to compare irisin' s diagnostic and prognostic value and specificity value in myocardial infarction with known markers of cardiac injury such as creatine kinase-MB isoenzyme (CK-MB) and troponin 3) to evaluate irisin as an early necrosis biomarker 4) To evaluate irisin's sensitivity as a biomarker to detect minor myocardial necrosis after elective percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infraction (MI) or with coronary artery disease without myocardial infraction who need percutaneous coronary intervention

Exclusion Criteria:

* age < 20 years old
* diseases or medications that could affect cardiac muscle or skeletal muscle metabolism
* musculoskeletal injury of surgery 6 months prior to recruitment
* severe liver or kidney disease (creatinine clearance < 60ml/min/1.73m2) or liver or kidney transplantation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
changes from baseline in serum irisin measured by ELISA | baseline and 6 hours or 24 hours

SECONDARY OUTCOMES:
changes from baseline in troponin | baseline and 6 hours or 24 hours
changes from baseline in serum lactate dehydrogenase | baseline and 6 hours or 24 hours
changes from baseline in serum creatine kinase | baseline and 6 hours or 24 hours
changes from baseline in serum creatine kinase-MB isoenzyme | baseline and 6 hours or 24 hours
changes from baseline in serum follistatin | baseline and 6 hours or 24 hours
changes from baseline in serum follistatin-like protein 3 (FSTL-3) | baseline and 6 hours or 24 hours
changes from baseline in serum Activin A | baseline and 6 hours or 24 hours
changes from baseline in serum Activin B | baseline and 6 hours or 24 hours
changes from baseline in serum insulin growth factor 1 (IGF1) | baseline and 6 hours or 24 hours
changes from baseline in serum insulin growth factor binding protein 3 (IGFBP3) | baseline and 6 hours or 24 hours
changes from baseline in serum insulin growth factor binding protein 4 (IGFBP4) | baseline and 6 hours or 24 hours
changes from baseline in serum pico pregnancy-associated plasma protein A (PAPP-A) | baseline and 6 hours or 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios D Anastasilakis, PhD, Principal Investigator — 424 General Military Hospital
Locations (1):
- 424 General Military Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Bostrom P, Wu J, Jedrychowski MP, Korde A, Ye L, Lo JC, Rasbach KA, Bostrom EA, Choi JH, Long JZ, Kajimura S, Zingaretti MC, Vind BF, Tu H, Cinti S, Hojlund K, Gygi SP, Spiegelman BM. A PGC1-alpha-dependent myokine that drives brown-fat-like development of white fat and thermogenesis. Nature. 2012 Jan 11;481(7382):463-8. doi: 10.1038/nature10777. PMID 22237023
- [Background] Stengel A, Hofmann T, Goebel-Stengel M, Elbelt U, Kobelt P, Klapp BF. Circulating levels of irisin in patients with anorexia nervosa and different stages of obesity--correlation with body mass index. Peptides. 2013 Jan;39:125-30. doi: 10.1016/j.peptides.2012.11.014. Epub 2012 Dec 3. PMID 23219488
- [Background] Huh JY, Panagiotou G, Mougios V, Brinkoetter M, Vamvini MT, Schneider BE, Mantzoros CS. FNDC5 and irisin in humans: I. Predictors of circulating concentrations in serum and plasma and II. mRNA expression and circulating concentrations in response to weight loss and exercise. Metabolism. 2012 Dec;61(12):1725-38. doi: 10.1016/j.metabol.2012.09.002. Epub 2012 Sep 25. PMID 23018146
- [Background] Aydin S, Kuloglu T, Aydin S, Eren MN, Celik A, Yilmaz M, Kalayci M, Sahin I, Gungor O, Gurel A, Ogeturk M, Dabak O. Cardiac, skeletal muscle and serum irisin responses to with or without water exercise in young and old male rats: cardiac muscle produces more irisin than skeletal muscle. Peptides. 2014 Feb;52:68-73. doi: 10.1016/j.peptides.2013.11.024. Epub 2013 Dec 15. PMID 24345335
- [Background] Kuloglu T, Aydin S, Eren MN, Yilmaz M, Sahin I, Kalayci M, Sarman E, Kaya N, Yilmaz OF, Turk A, Aydin Y, Yalcin MH, Uras N, Gurel A, Ilhan S, Gul E, Aydin S. Irisin: a potentially candidate marker for myocardial infarction. Peptides. 2014 May;55:85-91. doi: 10.1016/j.peptides.2014.02.008. Epub 2014 Feb 24. PMID 24576483
- [Background] Aydin S, Aydin S, Kobat MA, Kalayci M, Eren MN, Yilmaz M, Kuloglu T, Gul E, Secen O, Alatas OD, Baydas A. Decreased saliva/serum irisin concentrations in the acute myocardial infarction promising for being a new candidate biomarker for diagnosis of this pathology. Peptides. 2014 Jun;56:141-5. doi: 10.1016/j.peptides.2014.04.002. Epub 2014 Apr 18. PMID 24747283
- [Background] Aronis KN, Moreno M, Polyzos SA, Moreno-Navarrete JM, Ricart W, Delgado E, de la Hera J, Sahin-Efe A, Chamberland JP, Berman R, Spiro A 3rd, Vokonas P, Fernandez-Real JM, Mantzoros CS. Circulating irisin levels and coronary heart disease: association with future acute coronary syndrome and major adverse cardiovascular events. Int J Obes (Lond). 2015 Jan;39(1):156-61. doi: 10.1038/ijo.2014.101. Epub 2013 Jun 11. PMID 24916788